CLINICAL TRIAL: NCT06682130
Title: A Prospective Study of Glofitamab Bridging Autologous Peripheral Blood Stem Cell Transplantation for Patients With Relapsed and Refractory Diffuse Large B Cell Lymphoma.
Brief Title: Glofitamab Bridging ASCT for Patients With Relapsed or Refractory DLBCL
Acronym: ASCT DLBCL
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024378
Record Dates: First submitted 2024-11-07; First posted 2024-11-12 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Diffuse Large B-cell Lymphoma(DLBCL)
Keywords: Glofitamab; autologous stem cell transplantation
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Glofitamab bridging ASCT Regimen (Experimental): After at least second-line treatment, patients will be divided into three groups based on their disease status: Group A includes patients with partial response (PR) or ctDNA positivity who plan to receive ASCT or Glofitamab (specification: 10 mg per tube; dosage: 2.5 mg on day 8) as a bridge to ASCT; Group B includes patients with complete response (CR) and ctDNA negativity who will proceed directly to ASCT; Group C includes patients with stable or progressive disease (SD/PD) who will be assessed after two cycles of Glofitamab (Specification: 10mg per tube;Dosage: cycle 1: 2.5mg d8；10mg d15；cycle 2: 30mg d21). Those achieving PR will undergo ASCT, those with CR can choose ASCT or continue Glofitamab, and those with SD/PD will be removed from the group.
  Interventions: Drug: Group A：Patients with PR or ctDNA positivity after salvage treatment; Procedure: Group B: Patients with CR and ctDNA negative after salvage treatment; Drug: Group C: Patients with SD/PD after posterior treatment

INTERVENTIONS:
Drug: Group A：Patients with PR or ctDNA positivity after salvage treatment — 1. Immunotargeted therapy
     * Ottuzumab introvenous infusion, 1000mg day1;
     * Glofitamab introvenous infusion Group A: 2.5mg day8
  2. Autologous stem cell transplantation SEAM regimen
     * Simustine 250mg/m2 orally, day1
     * Etoposide 200mg/m2 intravenous infusion, day2-5
     * Cytarabine 400mg/m2 intravenous infusion, day2-5
     * Metformin 140mg/m2 intravenous infusion, day6; Patients in Group A who intend to receive Glofitamab+ASCT will receive Glofitamab 2.5mg on day8 and start ASCT pretreatment on day15.
Procedure: Group B: Patients with CR and ctDNA negative after salvage treatment — Group B patients initiated ASCT treatment directly after evaluating the efficacy of salvage treatment
Drug: Group C: Patients with SD/PD after posterior treatment — 1. Immunotargeted therapy
     * Ottuzumab introvenous infusion, 1000mg day1;
     * Glofitamab introvenous infusion Group C: cycle1 2.5mg day8, 10mg day15 cycle2 30mg day21
  2. Autologous stem cell transplantation SEAM regimen
     * Simustine 250mg/m2 orally, day1
     * Etoposide 200mg/m2 intravenous infusion, day2-5
     * Cytarabine 400mg/m2 intravenous infusion, day2-5
     * Metformin 140mg/m2 intravenous infusion, day6;
  After two treatment cycles with Glofitamab, patients in group C had a PET-CT to assess efficacy. Those with partial remission proceeded to ASCT consolidation, those with complete remission chose between ASCT or Glofitamab maintenance, and those with stable disease or progressive disease exited the trial.

SUMMARY:
The objective of this study is to evaluate the efficacy and safety of the Glofitamab bridging ASCT regimen in patients with relapsed/refractory (R/R) diffuse large B-cell lymphoma (DLBCL) and to provide better clinical benefits to these patients.

DETAILED DESCRIPTION:
This study seeks to include patients aged 18 to 70 years with relapsed or refractory diffuse large B-cell lymphoma (R/R DLBCL) who have undergone at least a second-line systemic treatment, excluding those with prior resistance to Glofitamab. Based on their disease status following the second-line treatment, participants will be categorized into three groups: A, B, and C. Group A will consist of patients who exhibit partial response (PR) or are circulating tumor DNA (ctDNA) positive after second-line treatment and are planning to undergo autologous stem cell transplantation (ASCT) or Glofitamab as a bridging therapy to ASCT. Group B will include patients who achieve complete response (CR) and are ctDNA negative post-second-line treatment, and they will receive ASCT as consolidation therapy. Patients in Group B who achieved CR and were ctDNA negative following second-line treatment will proceed directly to ASCT consolidation therapy. In Group C, patients who exhibited stable disease (SD) or progressive disease (PD) after second-line treatment were reassessed following two cycles of Glofitamab. Those who attained PR subsequently underwent ASCT consolidation therapy, whereas patients achieving CR had the option to either undergo ASCT or continue with Glofitamab maintenance therapy. Patients with SD or PD were excluded from the study. Patients exhibiting SD or PD were excluded from the cohort. Individuals who have successfully undergone autologous transplantation and subsequent maintenance therapy with Glofitamab will be monitored for assessments of efficacy and survival outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with diffuse large B-cell lymphoma (DLBCL) confirmed by histopathology/cytology using the 2022 World Health Organization (WHO) Classification of Diseases;
2. Patients with R/R DLBCL who have received at least two lines of systemic treatment;
3. Age range: 18-70 years old, male or female not limited;
4. When the disease recurs or is difficult to treat, there are assessable lesions (lymph node diameter ≥ 1.0cm; or skin lesions assessable by physical examination);
5. Expected lifespan>3 months;
6. No previous transplantation treatment has been performed;
7. ECOG score 0-1 points;
8. Appropriate organ function:

   Cardiac function: ejection fraction ≥ 50%, asymptomatic arrhythmia; Liver function: alanine aminotransferase and aspartate aminotransferase ≤ 2 times the upper limit of normal, total bilirubin<2 times the upper limit of normal; Renal function: serum creatinine clearance rate ≥ 80 mL/min, creatinine<160 umol/l; Pulmonary function: Without oxygen inhalation, SPO2>90%, FEV1, FVC, and DLCO ≥ 50% predicted values;
9. Adequate bone marrow reserve is defined as:

   Hemoglobin ≥ 9g/dL, Platelet count ≥ 70 × 10 ^ 9/L, The absolute value of neutrophils is ≥ 1.0 × 10 ^ 9/L, If accompanied by bone marrow invasion, platelet count ≥ 50 × 10 ^ 9/L, absolute neutrophil count ≥ 0.75 × 10 ^ 9/L, The number of CD34+cells is ≥ 2.0 × 109/kg.
10. The patient has the ability to understand and is willing to provide written informed consent.
11. Subjects with fertility or potential for fertility must be willing to undergo contraception from the date of registration in this study until the study follow-up period.

Exclusion Criteria:

-1) Previously underwent autologous hematopoietic stem cell transplantation; 2) HIV infection and/or active hepatitis B or C; 3) Uncontrolled active infections; 4) Severe liver and kidney dysfunction (alanine aminotransferase, bilirubin, creatinine>3 times the upper limit of normal); 5) Existence of organic heart disease or severe arrhythmia, leading to clinical symptoms or abnormal heart function (NYHA functional class ≥ 2); 6) Simultaneously present other tumors that require treatment or intervention; 7) Previous or current history of vascular embolism; 8) Pregnant or lactating women; 9) In a state of severe immune suppression; 10) Other psychological conditions that hinder patients from participating in research or signing informed consent forms.

11) According to the researcher's assessment, it is unlikely that the subjects will complete all the required study visits or procedures, including follow-up visits, or meet the requirements for participation in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-11-10 (Actual); Primary Completion 2027-11-10 (Estimated); Study Completion 2029-11-10 (Estimated)

PRIMARY OUTCOMES:
Complete remission rate(CRR) | At the end of 3 months after ASCT
  The rate of patients who achieved CR after treatment with Glofitamab bridging ASCT Regimen

SECONDARY OUTCOMES:
Main adverse reactions | Start from the first day of Immunotargeted therapy to 1 month after treatment with Glofitamab bridging ASCT Regimen
  The safety and tolerability of the therapeutic regimen measured by the major adverse events.
Overall response rate(ORR) | At the end of 3 months after ASCT.
  The rate of patients who achieved CR or PR after treatment with Glofitamab bridging ASCT Regimen
2-year progression-free survival(PFS) | From enrollment to 2 year after the treatment of last patient
  PFS will be assessed from the first day of Immunotargeted therapy to date of progression, relapse, death or end of follow-up.
2-year overall survival(OS) | From enrollment to 2 year after the treatment of last patient
  OS will be assessed from the first day of Immunotargeted therapy to date of death or end of follow-up.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No